CLINICAL TRIAL: NCT06441916
Title: A Single Dose, Randomized, Open-label, Two-treatment, Four-period, Two-sequence, Replicate Crossover Bioequivalence Study of Generic Dabigatran Etexilate Capsules 150 mg and Reference Product (Pradaxa®) in Healthy Thai Volunteers Under Fasting Conditions and Under Pre-treatment With a Proton Pump Inhibitor
Brief Title: Bioequivalence Study of Dabigatran Etexilate Capsules 150 mg in Healthy Thai Volunteers Under Fasting Conditions
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: International Bio service (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BE24-008
Record Dates: First submitted 2024-05-26; First posted 2024-06-04 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-04

CONDITIONS: Healthy Volunteer; Dabigatran; Bioequivalence Study
MeSH Terms: interventions — Dabigatran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dabigatran Etexilate Capsules 150 mg (Experimental): Each capsule contains Dabigatran Etexilate 150 mg
  Interventions: Drug: Dabigatran Etexilate Capsules 150 mg
- Pradaxa® (Active Comparator): Dabigatran Etexilate
  Interventions: Drug: Dabigatran Etexilate Capsules 150 mg

INTERVENTIONS:
Drug: Dabigatran Etexilate Capsules 150 mg — Dabigatran Etexilate
  Other Names: Dabigatran

SUMMARY:
The bioequivalence of Dabigatran Etexilate Capsules 150 mg to Boehringer Ingelheim's Pradaxa® will be assessed by a statistical comparison of various pharmacokinetic parameters derived from the plasma concentration-time curves of free dabigatran and total dabigatran.

DETAILED DESCRIPTION:
Bioequivalence study is a research study that needs to compare the rate and extent to which the active substance or active moiety is absorbed from a pharmaceutical dosage form between innovator or reference product and test product when given in healthy subjects at the same dose and strength. The acceptance criteria in bioequivalence study will be done by comparing the pharmacokinetic parameters including maximal plasma concentration (Cmax) time at which the maximum plasma concentration occurs (Tmax) and area under the plasma concentration curve (AUC) either area under the plasma concentration curve from administration to last observed concentration at time t (AUC0-tlast) or area under the plasma concentration curve extrapolated to infinite time (AUC0-∞). Those parameters should be calculated only from the plasma concentration and time curve but cannot use other data obtained from in vitro study. By this reason, it is necessary to conduct the study in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy Thai male or female subjects between the ages of 18 to 55 years. Subject must meet age requirements at the time of signing the initial informed consent and at the dosing day in Period 1.
* Body mass index between 18.5 to 30.0 kg/m2
* Normal laboratory values, including vital signs and physical examination, for all parameters in clinical laboratory tests at screening. Any abnormalities from the normal or reference range will be carefully considered clinically relevant by the physician as individual cases, documented in study files prior to enrolling the subject in this study
* Non-smoker and non-consumer of nicotine containing products. Non-smoker or non-consumer of nicotine containing products means any subject who has never smoked/consumed or stopped for at least 90 days.
* Non-pregnant woman (negative pregnancy test) and not currently breast feeding.
* Female subjects abstain from either hormonal methods of contraception (including oral or transdermal contraceptives, injectable progesterone, progestin subdermal implants, progesterone-releasing IUDs, postcoital contraceptive methods) or hormone replacement therapy for at least 28 days prior to check-in in Period 1. Injectable contraceptives e.g. Depo-Provera® will be discontinued at least 6 months prior to check-in in Period 1. Subjects agree to use acceptable non-hormonal contraceptive methods such as condom, diaphragm, foams, jellies, or abstinence for at least 14 days prior to check-in in Period 1 until 7 days after the end of study in Period 4. Female subjects of non-childbearing potential must meet at least one of the following criteria prior to check-in in Period 1:
* Postmenopausal for at least 1 year or
* Surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy) at least 6 months
* Male subjects who are willing or able to use effective contraceptive e.g. condom or abstinence after check-in in Period 1 until 7 days after the end of study in Period 4.
* Able to understand and voluntarily given written informed consent (signed and dated) by the subject prior to participating in this study.
* Adequate venous access in both arms for the collection of a number of samples during the study.

Exclusion Criteria:

* History of hypersensitivity to dabigatran or dabigatran etexilate or to any of the excipients of product
* History or evidence of clinically significant renal, hepatic, gastrointestinal, hematological (e.g. anemia), endocrine (e.g. hyper-/hypothyroid, diabetes), pulmonary or respiratory (e.g. asthma), cardiovascular (e.g. hyper-/hypotension), psychiatric (e.g. depression), neurologic (e.g. convulsant), allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing) or any significant ongoing chronic medical illness. Have high risk for coronavirus infection based on risk assessment questionnaire or diagnosed as confirmed case of COVID-19.
* History about administration of COVID-19 vaccine within 30 days prior to check-in in each Period.
* Have eGFR (CKD-EPI) < 50 mL/min/1.73 m2 based on serum creatinine results, at the screening laboratory test or during enrollment.
* History or evidence of haemorrhagic manifestations, patients with a bleeding diathesis or patients with spontaneous or pharmacological impairment of haemostasis.
* History or evidence of organ lesions at risk of clinically significant bleeding, including haemorrhagic stroke within the last 6 months.
* History or evidence of surgery for prosthetic heart valve replacement.
* History or evidence of surgery for knee or hip replacement.
* History or evidence of venous thromboembolic events, deep vein thrombosis or pulmonary embolism.
* History or evidence of stroke.
* History or evidence of atrial fibrillation.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Any condition possibly affecting drug absorption e.g. gastrectomy, enterectomy, gastritis or duodenal or gastric ulceration other than appendectomy.
* History of diarrhea or vomiting within 24 hours prior to check-in in each period.
* History of problems with swallowing tablet or capsule.
* History or evidence of drug addict or investigation with urine sample shows a positive test for drug of abuse (morphine, marijuana or methamphetamine).
* 12-lead ECG demonstrating QTc > 450 msec, a QRS interval > 120 msec or with an abnormality considered clinically significant at screening. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG will be repeated two more times and the average of the three QTc or QRS values will be used to determine the subject's eligibility.
* Investigation with blood sample shows positive test for HBsAg.
* Abnormal liver function, ≥1.5 times of upper normal limit of reference range for ALT, AST or bilirubin levels at screening laboratory test. History or evidence of alcoholism or harmful use of alcohol (less than 2 years) i.e., alcohol consumption of more than 14 standard drinks per week for men and 7 standard drinks per week for women (A standard drink is defined as 360 mL of beer or 150 mL of wine or 45 mL of 40% distilled spirits, such as rum, whisky, brandy etc.).
* History or evidence of alcohol consumption or alcohol-containing products and cannot abstain for at least 48 hours prior to check-in and continued for entire duration of the study or alcohol breath test shows positive result In case of alcohol breath test result represents the alcohol concentration range of

  1 - 10 mg% BAC and the physician carefully considers that the value came from other reasons, not from the alcohol drinking behavior of subjects, the test will be repeated two times separately, not more than 10 minutes. The result of the last time should be used for subject's eligibility which must be 0 mg%BAC.
* History or evidence of habitual consume of any caffeine- or xanthine-containing products e.g. tea, coffee, chocolate, colas etc. and cannot abstain for at least 72 hours prior to check-in and continued for entire duration of the study.
* Consume or drink juice of grapefruit or orange or pomelo or its supplement/ containing products and cannot abstain for at least 7 days prior to check-in and continued for entire duration of the study.
* Use of prescription or nonprescription drugs (e.g. paracetamol, amiodarone, verapamil, quinidine, ketoconazole, dronedarone, ticagrelor, clarithromycin, other anticoagulants, NSAIDs, selective serotonin reuptake inhibitors, selective serotonin norepinephrine reuptake inhibitors, fibrinolytic agents and etc.), herbal medications or supplements (e.g. St. John's wort), vitamins or mineral (e.g. iron) or dietary supplements within 14 days prior to check-in in Period 1 and continued for entire duration of the study
* Participated in other clinical trials within 90 days prior to check-in in Period 1 (except for the subjects who drop out or withdrawn from the previous study prior to Period 1 dosing) or still participates in the clinical trial or participates in other clinical trials during enrollment in this study
* Blood donation or blood loss ≥ 1 unit (1 unit is equal to 350-450 mL of blood) within 90 days prior to check-in in Period 1 or during enrollment.
* Subjects with poor venous access or intolerant to venipuncture.
* Unwilling or unable to comply with schedule visit, treatment plan and other study procedures until end of study.
* Inability to communicate well (i.e. language problem, poor mental development, psychiatric illness or poor cerebral function) that may impair the ability to provide written informed consent or cooperate with clinical team.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-25 (Estimated); Primary Completion 2024-10-08 (Estimated); Study Completion 2024-11-07 (Estimated)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) of Dabigatran | Through 48 Hours Post Dose
  Maximum measured plasma concentration over the time span specified.
Plasma Area Under the Curve AUC(0 to 48hr, AUC0-∞ | Through 48 Hours Post Dose
  The area under the plasma concentration versus time curve.

CONTACTS AND LOCATIONS:
Overall Officials: Porranee Puranajoti, Ph. D, Principal Investigator — International Bio Service Co., Ltd.